CLINICAL TRIAL: NCT05337514
Title: Voice-Activated Technology to Improve Mobility in Multimorbid, Frail, Homebound Older Adults: EngAGEing Older Adult-Care Partner Dyads
Brief Title: Voice-Activated Technology to Improve Mobility in Multimorbid, Frail, Homebound Older Adults (EngAGE)
Acronym: EngAGE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Rush University (Other); National Opinion Research Center (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB21-1556; P50MD017349 (NIH)
Record Dates: First submitted 2022-04-13; First posted 2022-04-20 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Frailty
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EngAGE (Experimental): Older adult subjects will receive an Alexa Echo Show that runs an exercise app called EngAGE.
  Interventions: Behavioral: Enhanced Engagement
- Physical Exercise Handouts (Active Comparator): Older adults subjects will receive a paper booklet containing exercise instructions.
  Interventions: Behavioral: Standard Engagement

INTERVENTIONS:
Behavioral: Enhanced Engagement — EngAGE will allow care partners send older adults encouragement which will be read aloud to the older adult through the EngAGE app.
  Arms: EngAGE
Behavioral: Standard Engagement — Care partners can encourage their older adult partner using traditional / existing communication mechanisms.
  Arms: Physical Exercise Handouts

SUMMARY:
The purpose of this study is to test the efficacy of EngAGE (an interactive, voice-activated app) vs usual care on improving older adult physical and social function.

DETAILED DESCRIPTION:
Physical activity is essential for all age groups, across all comorbidities and geriatric syndromes; it has been described as the 'ideal' intervention for aging. Increasing physical activity among homebound, multimorbid, African American (AA) older adults (OAs) requires a shift in interventions to target the older adult-care partner (CP) pair (dyad) and to test innovative vehicles for remote intervention delivery. Our research goal is to create an evidence-based intervention that leverages technology to reach multimorbid OA-CP dyads in the home, promotes long-term mobility and social engagement among those least able to access community resources, and empowers informal care partners with tools. We developed a socially-motivated exercise tool for multimorbid OA-CP dyads called EngAGE that leverages voice-activated technology. We propose to conduct a 6-month, randomized, in-home trial of EngAGE (intervention) versus paper exercise handouts (usual care) in 124 multimorbid, homebound, AA OA-CP dyads recruited from 2 hospital systems and the community. Our overall hypothesis is that EngAGE will improve both physical and social function of older adults.

All OA subjects will undergo an in-home baseline visit where we will collect data about physical function, social function, activity and frailty. OA-CP dyads will be randomized (1:1) to a physical activity intervention: either EngAGE or usual care. All subjects will be asked to complete exercises 3-6 times per week. Care Partners will be instructed to encourage their Older Adult partner to perform physical activities on a regular basis. There is a two week Run-In Period to troubleshoot the EngAGE app and acclimate the OA subjects to the study intervention. OA subjects will be monitored via phone visits on a monthly basis. In home study visits will take place at month 3 and month 6. Data about OA subject physical function, social function, activity and frailty will be collected at these visits.

ELIGIBILITY:
Inclusion Criteria:

* age greater than or equal to 60 years
* has at least 2 chronic conditions
* requires any assistance to leave the home (this may include requiring someone to drive, requiring the use of a cane or walker, or similar)
* can read 14 point font from a 2-foot distance on a tablet-sized screen
* can hear spoken voice from 2-foot distance
* SPPB score of less than or equal to 9 but greater than 3 on a 12-point scale to target moderate but not severe functional impairment.

Exclusion Criteria:

* reported history of moderate to advanced cognitive impairment;
* inability to stand unassisted;
* inability to understand English (because the intervention is currently only available in English);
* life expectancy less than 12 months or enrolled in Hospice;
* a medical condition making unsupervised physical activity potentially unsafe including: stroke within prior 12 months, acute myocardial infarction or unstable angina in the prior 6 months, uncontrolled arrhythmias, dissecting aortic aneurysm, acute endo/pericarditis, acute thromboembolism, acute or severe heart or respiratory failure, uncontrolled hypertension greater than 180/100, fracture or joint replacement within the prior 3 months, infections affecting one's general health condition, severe peripheral vascular disease.
* severe functional impairment as indicated by an SPPB score less than 3 (out of 12);
* baseline Montreal Cognitive Assessment of less than or equal to 18/30;
* inability to understand consent (teach back).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2022-10-26 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Timed Chair Stands | 6 months
  5 repeated chair stands

SECONDARY OUTCOMES:
Grip Strength | 6 months
  Dominant grip strength measured with a dynamometer, average of 3 attempts
Loneliness | 6 months
  Measured with the 9-item UCLS loneliness scale
4 meter usual walk | 6 months
  Participants walk 4 meters 2 times at their usual pace, fastest of 2 attempts.
Static Balance Poses | 6 months
  Participants are asked to hold a side-by-side, semi-tandem and tandem balance pose each for 10 seconds.
Physical activity | 6 months
  Wrist accelerometers will be worn for 7 full days in the free living environment.

CONTACTS AND LOCATIONS:
Overall Officials: Megan Huisingh-Scheetz, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No